CLINICAL TRIAL: NCT05016128
Title: Second Affiliated Hospital Zhejiang University School of Medicine
Brief Title: Intraoperative S-ketamine to Prevent Postoperative Hyperalgesia in Patients Undergoing Video-assisted Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0442
Record Dates: First submitted 2021-08-09; First posted 2021-08-23 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Hyperalgesia
MeSH Terms: interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine (Experimental): a 0.25 mg/kg bolus and 0.125 mg/kg/h via intravenous infusion during surgery
  Interventions: Drug: S-ketamine
- Saline (Placebo Comparator): a 0.25 mg/kg bolus and 0.125 mg/kg/h via intravenous infusion during surgery
  Interventions: Drug: saline

INTERVENTIONS:
Drug: S-ketamine — S-ketamine is used for preventing postoperative hyperalgesia,thus reducing the patient's acute postoperative pain
  Other Names: esketamine
  Arms: S-ketamine
Drug: saline — saline is used for control
  Other Names: 0.9%saline
  Arms: Saline

SUMMARY:
Postoperative hyperalgesia (POH) is a paradoxical clinical state of increased sensation of pain or increased sensitivity to non-painful stimuli at the site of surgery or at a surrounding area that was not directly injured. Opioid-induced hyperalgesia (OIH) and nociceptive-induced hyperalgesia (NIH) are the two main causes of POH.N-methyl-D-aspartate receptor (NMDAR) activation plays a central role in the development of POH.S-ketamine，which is a NMDA-receptor antagonist,has been on the market in china since 2019.The aim of this study is to evaluate the effects of S-ketamine on POH and chronic postoperative pain after video-assisted thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class I-III.
* elective single-port video-assisted thoracic surgery under general

Exclusion Criteria:

* a history of thoracic surgery
* a history of chronic pain
* ongoing pain treatment
* opioid drug or alcohol abuse
* a history of allergy to anesthetics
* obesity (body mass index [BMI] >30 kg/m2 )
* pregnancy
* psychiatric disorders
* neurological disease
* severe diabetes
* renal or hepatic insufficiency
* uncontrolled hypertension, or arrhythmia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
the mechanical pain threshold around the incision | Day1 after surgery
  the mechanical pain threshold was assessed by using 10 calibrated (4-300 g mm-2 ) hand-held Von Frey filaments (North Coast Medical Inc.USA)around the skin incision.The per pain threshold was defined as the smallest force (g mm-2 ) necessary to bend a von Frey hair, and perceived by the patient as three consecutive painful stimuli with approximately 10 s elapsing between two successive stimuli. The mechanical pain threshold was recorded as the mean of 6 measurements at 2 cm vertically above and below the middle and bilateral edges of the incision.

SECONDARY OUTCOMES:
the mechanical pain threshold on the forearm | the day before surgery
  the mechanical pain threshold was assessed by using 10 calibrated (4-300 g mm-2 )hand-held Von Frey filaments (North Coast Medical Inc. USA)on the nondominant inner forearm The per pain threshold was defined as the smallest force (g mm-2 ) necessary to bend a von Frey hair, and perceived by the patient as three consecutive painful stimuli with approximately 10 s elapsing between two successive stimuli. The mechanical pain threshold was recorded as the mean of 3 measurements at 3, 6, and 9 cm distal to the middle of the antecubital crease
the mechanical pain threshold | Day1 after surgery
  the mechanical pain threshold was assessed by using 10 calibrated (4-300 g mm-2 )hand-held Von Frey filaments (North Coast Medical Inc.USA)on the nondominant inner forearm The per pain threshold was defined as the smallest force (g mm-2 ) necessary to bend a von Frey hair, and perceived by the patient as three consecutive painful stimuli with approximately 10 s elapsing between two successive stimuli. The mechanical pain threshold was recorded as the mean of 3 measurements at 3, 6, and 9 cm distal to the middle of the antecubital crease .
the mechanical pain threshold | Day2 after surgery
  the mechanical pain threshold was assessed by using 10 calibrated (4-300 g mm-2 )hand-held Von Frey filaments (North Coast Medical Inc.USA)on the nondominant inner forearm The per pain threshold was defined as the smallest force (g mm-2 ) necessary to bend a von Frey hair, and perceived by the patient as three consecutive painful stimuli with approximately 10 s elapsing between two successive stimuli. The mechanical pain threshold was recorded as the mean of 3 measurements at 3, 6, and 9 cm distal to the middle of the antecubital crease .
the mechanical pain threshold around the incision | Day2 after surgery
  the mechanical pain threshold was assessed by using 10 calibrated (4-300 g mm-2 ) hand-held Von Frey filaments (North Coast Medical Inc. USA)around the skin incision.The per pain threshold was defined as the smallest force (g mm-2 ) necessary to bend a von Frey hair, and perceived by the patient as three consecutive painful stimuli with approximately 10 s elapsing between two successive stimuli. The mechanical pain threshold was recorded as the mean of 6 measurements at 2 cm vertically above and below the middle and bilateral edges of the incision.
postoperative pain scores | up to day2 after surgery
  postoperative pain scores was assessed by using numeric rating scales(0-10,0 means"better ',10 means "worst") at 6 time points:1 hours,3 hours,6 hours, 12 hours,24 hours, and 48 hours after the operation. The worst pain score during each interval was recorded.
Anxiety scale scores | up to day2 after surgery
  Anxiety scale scores was assessed by Hamilton Anxiety Scale at three time points:the day before surgery, day1 after surgery and day2 after surgery.
  If the total score exceeds 29 points, it may be severe anxiety. If the score exceeds 21 points, there must be obvious anxiety. If the score exceeds 14, there must be anxiety. If it exceeds 7 points, there may be anxiety. If it is less than 6, the patient has no anxiety symptoms.
Depression scale scores | up to day2 after surgery
  Depression scale scores was assessed by Hamilton Depression Scale at three time points:the day before surgery, day1 after surgery and day2 after surgery.
  The total score is less than 7 points, normal; 7-17 points, there may be depression. 17-24 points, there must be depression, more than 24 points, severe depression.
The hyperalgesic area around the incision | up to day2 after surgery
  The hyperalgesic area around the surgical incision was measured by the von Frey filament that in postoperative pain threshold testing evoked pain on the opposite side. Stimulation was started far from the surgical incision and moved toward the incision in 0.5 cm steps until the patient reported a distinct change in pain perception. The first point at which the patient reported a more painful, sore or sharp feeling was marked, and the distance to the incision was measured . Finally, we calculated the incidence and extension of peri-incisional mechanical hyperalgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated Hospital School of Medicine,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No